CLINICAL TRIAL: NCT03343535
Title: Trial to Evaluate the Safety and Effectiveness of the Portable Organ Care System (OCS™) Lung System for Recruiting, Preserving and Assessing Non-Ideal Donor Lungs for Transplantation
Brief Title: OCS Lung System EXPAND II Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment in EXPAND II was stopped June 24, 2019 as a result of the FDA approval for the EXPAND indication. Therefore, no additional sites or subjects were enrolled after that time.
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCS-LUN-012017
Record Dates: First submitted 2017-11-08; First posted 2017-11-17 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-11

CONDITIONS: Lung Transplantation
Keywords: portable ex-vivo lung perfusion; breathing lung transplant; portable OCS Lung System

STUDY DESIGN:
Intervention Model Description: OCS Lung System
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- OCS Preservation (Experimental)
  Interventions: Device: OCS Lung Preservation

INTERVENTIONS:
Device: OCS Lung Preservation — OCS Lung Preservation
  Other Names: OCS Lung Transplant

SUMMARY:
To evaluate the safety and effectiveness of the OCS™ Lung System to recruit, preserve and assess non-ideal donor lungs that may not meet current standard donor lung acceptance criteria for transplantation.

DETAILED DESCRIPTION:
Inclusion

At least one of the following:

* Donor PaO2/FiO2 ≤ 300 mmHg at the time of the offer; or
* Expected cross-clamp time > 6 hours for the second lung; or
* Donor after Cardiac Death (DCD donor); or
* Donor age ≥ 55 years old

ELIGIBILITY:
Inclusion Criteria:

* Male or female primary double lung transplant candidate
* Age ≥ 18 years old
* Signed: 1) written informed consent document and 2) authorization to use and disclose protected health information

Exclusion Criteria:

* Prior solid organ or bone marrow transplant
* Single lung recipient
* Chronic use of hemodialysis or renal replacement therapy for diagnosis of chronic renal dysfunction requiring dialysis
* Participant in any other clinical or investigational trials/programs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2022-07-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - UCLA Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Nebraska, Omaha, Nebraska
  - Duke University Medical Center, Durham, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Houston Methodist, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 51 Donor Lungs were instrumented on OCS Lung and 46 Donor Lungs were accepted and transplanted on study.
Pre-assignment Details: Enrollment was stopped as a result of the FDA Approval of OCS Lung for the EXPAND indication.
Period: Overall Study
Arm/Group | OCS Preservation
Started (Donor Lungs Transplanted) | 46
Completed (36-month follow-up completed) | 32
Not Completed | 14
Not completed — Lost to Follow-up | 1
Not completed — Subject Discontinued Due to Re-transplant | 1
Not completed — Death | 12

BASELINE CHARACTERISTICS:
Arm/Group | OCS Preservation
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] — Recipient Age (years)
  years | 54.5 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Recipient Gender
  Participants
    Female | 19
    Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 36
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Patient Survival
Description: Patient survival at Day-30 post-transplantation or initial hospital discharge post-transplantation, whichever occurs later.
Time Frame: 30 days post-transplantation or initial hospital discharge post-transplantation, a mean of 41.5 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | OCS Preservation
Number analyzed (Participants) | 46
Participants | 40

2. Primary Outcome: Donor Lung Utilization Rate
Description: Donor lung utilization rate, defined as the number of donated lungs instrumented on OCS™ that meet inclusion/exclusion criteria for the trial and acceptance criteria for transplantation after OCS™ Lung assessment divided by the total eligible donor lungs instrumented on the OCS™ Lung System.
Time Frame: Immediately at Transplantation
Population: 51 eligible donor lungs were instrumented on OCS. 46 donor lungs were accepted after perfusion and transplanted into recipients.
Measure: Count of Units; unit: Lungs Instrumented on OCS
Units Other Than Participants: Lungs Instrumented on OCS
Arm/Group | OCS Preservation
Number analyzed (Participants) | 46
Number analyzed (Lungs Instrumented on OCS) | 51
Lungs Instrumented on OCS | 46

3. Secondary Outcome: Primary Graft Dysfunction Grade 3
Description: Number of Participants with Primary Graft Dysfunction Grade 3 at T72 hours
Time Frame: 72 hours post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | OCS Preservation
Number analyzed (Participants) | 46
Participants | 7

4. Other Pre Specified Outcome: Number of Lung Graft-related Serious Adverse Events
Description: Number of lung graft-related serious adverse events through the 30-day follow-up or until initial hospital admission (if longer than 30 days) after transplantation per subject.
Time Frame: 30 days post-transplantation or initial hospital discharge post-transplantation, a mean of 41.5 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | OCS Preservation
Number analyzed (Participants) | 46
Participants | 16

ADVERSE EVENTS:
Time Frame: Lung graft related SAEs (LGRSAEs) data was collected for transplanted recipients through 30-days post-transplant or through the initial hospital stay, if longer than 30 days (a mean of 41.5 days post-transplant). All cause mortality is reported through 36-months post-transplant for all transplanted recipients.
Description: Non-serious adverse events were not captured as part of this study. Only lung graft related SAEs and deaths were captured through investigator assessment.
Arm/Group | OCS Preservation
All-Cause Mortality (participants affected / at risk) | 12/46
Serious Adverse Events (participants affected / at risk) | 16/46
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OCS Preservation (N=46)
Respiratory failure/protracted ventilation (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Major pulmonary-related infection (Infections and infestations) | 7 (8)
Bronchial anastomotic complication (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Biopsy-proven moderate or severe acute rejection (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site shall have right to publish results. To balance this right with TransMedics' (TM proprietary interests, site will submit manuscripts intended for publication for TM's review at least 30d prior to submission date. TM will complete its review within 30d of receipt. TM may request that site delete from its manuscripts any reference to TM confidential information and site shall promptly comply with such request. After 60d period, site will have right to publish manuscript, as amended by TM.

DOCUMENTS (2):
  • Study Protocol (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT03343535/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT03343535/SAP_001.pdf